CLINICAL TRIAL: NCT01559480
Title: A Prospective Double Blind Randomized Controlled Trial to Study the Effectiveness of a Desogestrel for the Treatment of Pelvic Pain or Dysmenorrhea in the Patients Undergone Conservative Surgery for Pelvic Endometriosis
Brief Title: Postoperative Desogestrel for Endometriosis Related Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R015532018
Record Dates: First submitted 2012-03-12; First posted 2012-03-21 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Endometriosis
Keywords: Endometriosis; Desogestrel; Placebo
MeSH Terms: conditions — Endometriosis | interventions — Desogestrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desogestrel (Active Comparator)
  Interventions: Drug: Desogestrel
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desogestrel — Desogestrel 75 mcg Takes 1 capsule before bedtime for 6 months
  Other Names: Cerazette
  Arms: Desogestrel
Drug: Placebo — Placebo capsule takes 1 capsule before bedtime for 6 months
  Arms: Placebo

SUMMARY:
Endometriosis is one of the most common disease in reproductive aged women.Surgical intervention has a significant symptoms relief. However, symptom recurrence is often after surgery. This study aims to determine the efficacy of Desogestrel compared with placebo in pain symptom of symptomatic endometriosis patient undergo conservative surgery . The primary outcome measurement is pain score at 6 months after surgery.

DETAILED DESCRIPTION:
After conservative surgery, the patients are randomized to Desogestrel and placebo groups. VAS pain score are compared after complete 6 months

ELIGIBILITY:
Inclusion Criteria:

* diagnoses endometriosis
* Plan conservative surgery
* initial pain score at least 5
* voluntary to be the participant of this study with inform consent
* No desired child bearing in 6 months

Exclusion Criteria:

* residual lesion after surgery which required further treatment
* cannot participate complete 6 months after surgery
* contraindication for Desogestrel, Paracetamol or Ponstan
* Pregnant

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Pain score | 6 months
  Pain score will be assessed by visual analog scale (0-10)

SECONDARY OUTCOMES:
Side effect compared between both group | 6 month
Patients satisfaction compare between both groups | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Prasong Tanmahasamut, M.D., Principal Investigator — Mahidol University
Locations (2):
- Thailand (2):
  - Faculty of medicine Siriraj hospital, Mahidol university, Bangkok Noi, Bangkok
  - Siriraj hospital Mahidol university, Bangkok Noi, Bangkok

REFERENCES:
- [Derived] Chen I, Kives S, Zakhari A, Nguyen DB, Goldberg HR, Choudhry AJ, Le AL, Kowalczewski E, Schroll JB. Progestagens for pain symptoms associated with endometriosis. Cochrane Database Syst Rev. 2025 Oct 9;10(10):CD002122. doi: 10.1002/14651858.CD002122.pub3. PMID 41065045